CLINICAL TRIAL: NCT00462176
Title: A Retrospective Follow-up of Patients After Laparoscopic Segmental Bowel Resection for Deep Infiltrating Colorectal Endometriosis
Brief Title: Laparoscopic Segmental Bowel Resection for Deep Infiltrating Colorectal Endometriosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Christel Meuleman, MD, University Hospitals Leuven, Leuven, Belgium
Other Study IDs: ML2818 - 20/02/2006 a
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Endometriosis
Keywords: colorectal endometriosis; deep infiltrating endometriosis; dysmenorroe; dyspareunia; quality of life
MeSH Terms: conditions — Endometriosis; Dyspareunia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The diagnosis of endometriosis was confirmed by histologic examination of resected lesions.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All women (n=45) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of the colorectal surgeon performing a bowel resection were selected retrospectively from the list of all patients (n=more than 400) operated at the Leuven University Fertility Centre (LUFc) between September 2004 and July 2006.
  Interventions: Procedure: multidisciplinary laparoscopy; Other: Questionnaires

INTERVENTIONS:
Procedure: multidisciplinary laparoscopy — Laparoscopic segmental bowel resection for deep infiltrating colorectal endometriosis performed by an experienced colorectal surgeon.
Other: Questionnaires — All 45 patients were asked to complete the Oxford Endometriosis Quality of Life questionnaire, a sexual activity questionnaire, visual analogue scales (VAS) for dysmenorroe, chronic pelvic pain and deep dyspareunia, and to answer questions about medication and fertility, to compare their status before surgery and at the moment of the evaluation (December 2008).

SUMMARY:
This study is executed to evaluate the outcome on quality of life, pain, sexuality, pregnancy rate and recurrence rate after a fertility sparing multidisciplinary CO2 laser laparoscopic radical excision of deep infiltrating colorectal endometriosis with a bowel resection.

DETAILED DESCRIPTION:
Patients

All women (n=45) who had undergone fertility sparing CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with bowel resection were selected retrospectively from the list of all patients (n=more than 500, of whom slightly more than 50% with endometriosis) operated at the Leuven University Fertility Centre (LUFc) between September 2004 and September 2006.

Questionnaires

All 45 patients were asked to complete the Oxford Endometriosis Quality of Life questionnaire (27), a sexual activity questionnaire (28), visual analogue scales (VAS) for dysmenorroe, chronic pelvic pain and deep dyspareunia, and to answer questions about medication and fertility, to compare their status before surgery and at the moment of the evaluation (December 2008).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from deep infiltrating endometriosis with colorectal extension
* Who had undergone CO2 laser laparoscopic radical excision of the endometriosis
* with bowel resection performed by the colorectal surgeon
* between September 2004 and July 2006.

Exclusion Criteria:

* Patients without bowel resection

Ages: 19 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All women (n=45) who had undergone CO2 laser laparoscopic radical excision of deep infiltrating endometriosis with active involvement of the colorectal surgeon performing a bowel resection were selected retrospectively from the list of all patients (n=more than 400) operated at the Leuven University Fertility Centre (LUFc) between September 2004 and July 2006.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2004-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Pain; Sexuality; Quality of life; Fertility rate; Complication rate; Recurrence rate | a median follow-up of 27 months (range 16 - 40 months) after surgery

SECONDARY OUTCOMES:
Economic life circumstances | a median follow-up of 27 months (range 16 - 40 months) after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christel LC Meuleman, MD, Principal Investigator — University Hospital Gasthuisberg, Leuven, Belgium; Thomas D'Hooghe, MD, PhD, Study Director — University Hospital Gasthuisberg, Leuven, Belgium
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium